CLINICAL TRIAL: NCT05741411
Title: Utilizing Mobile Health to Expedite Access to Specialty Care for Youth Presenting to the Emergency Department With Concussion at Highest Risk of Developing Persisting Symptoms
Brief Title: Facilitating Access to Specialty Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-019755; K23NS128275 (NIH)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Mild Traumatic Brain Injury; Concussion, Mild; Concussion, Severe; Concussion, Intermediate
Keywords: mobile health; emergency department; persistent post-concussion symptoms; remote patient monitoring
MeSH Terms: conditions — Brain Concussion; Emergencies

STUDY DESIGN:
Intervention Model Description: Single group intervention arm compared to historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concussed youth at risk for prolonged symptoms (Experimental)
  Interventions: Other: RPM-assisted specialist access

INTERVENTIONS:
Other: RPM-assisted specialist access — Participants will be prompted to report current symptoms and activity once a day via remote patient monitoring chat technology for up to 28 days following injury. Patients with either escalating or plateauing symptoms will be flagged, with an electronic alert sent via the electronic health record to a nurse navigator. The nurse navigator will have access to the symptom data and facilitate scheduling an in person or telehealth specialist visit as indicated. Symptoms will continue to be monitored through the 28-day acute study period with additional clinical visits occurring according to clinical need.

SUMMARY:
The goal of this hybrid implementation-effectiveness study is to evaluate the effectiveness (hastened recovery times) and feasibility (fidelity in connecting to concussion specialty care) of a novel mobile health intervention, designed to reduce disparities in access to specialty care through the use of remote patient monitoring (RPM) to facilitate care hand-off from the emergency department (ED) to concussion specialty care. Participants will report their symptoms and activity once daily through RPM chat technology that is linked to their electronic health record and prompts referral to specialty care.

ELIGIBILITY:
Inclusion Criteria for concussed subjects:

* Males and females age 13 - 18
* Present to the Children's Hospital of Philadelphia (CHOP) Emergency Department (ED) within 72 hours of head injury
* Meet criteria for concussion as defined by the most recent International Consensus Statement on Concussion
* Own a smartphone
* Meet criteria for moderate-to-high risk for Persistent Post-Concussion Symptoms according to 5P rule (score >3/12)

Exclusion Criteria for concussed subjects:

* Glasgow Coma Scale score <13
* Lower extremity trauma
* A prior concussion within 1 month
* Non-English speaking
* Admission to the hospital at the initial head injury visit
* Previously enrolled in the study
* Inability to complete study procedures.

Inclusion Criteria for parents:

* Child meets the study eligibility criteria

Exclusion Criteria for parents:

* Non-English speaking

Inclusion Criteria for providers:

* ED or specialty provider caring for at least one patient via the mobile Health (mHealth)-facilitated care handoff strategy

Exclusion Criteria for providers:

* Non-English speaking

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Persisting Post-Concussion Symptoms (PPCS, Primary Effectiveness) | 28 days from injury
  Persistence of at least 3 concussion-like symptoms above the pre-injury state beyond 28 days from injury, defined as a positive difference between patient-reported symptoms and the perceived pre-injury symptom rating
Percent of participants meeting referral criteria who interact with a specialty care provider (Fidelity, Primary Implementation) | 28 days from injury
  Among those participants who flag to see a specialist, at least 1 interaction with a specialty provider either in person or via telehealth during the acute study period

SECONDARY OUTCOMES:
Modeling of PPCS (Secondary Effectiveness) | 28 days from injury
  Multivariate logistic regression evaluating the effect on the incidence of PPCS of socio-demographic and neighborhood-level economic variables, including race, ethnicity, sex, insurance, mechanism of injury, and child opportunity index, as well as known factors associated with PPCS, including age, concussion history, and co-morbid conditions
Days until return to symptoms baseline (Secondary Effectiveness) | Up to 90 days from injury
  Number of days from injury whereby patient-reported symptoms meets pre-injury baseline levels
Days until clearance (Secondary Effectiveness) | Up to 90 days from injury
  Number of days from injury until patient is fully cleared for full activity by a medical provider
Days until return to school (Secondary Effectiveness) | Up to 90 days from injury
  Number of days from injury until patient is able to return to full time school without accommodations
Modeling of fidelity (Secondary Implementation) | 28 days from injury
  Multivariate logistic regression evaluating the effect on fidelity of socio-demographic and neighborhood-level economic variables, including race, ethnicity, sex, insurance, mechanism of injury, and child opportunity index
Patient-defined quantitative appropriateness (Secondary Implementation) | Within 1 year of completing study procedures
  Mean System Usability Score out of 100 with >=70 defined as acceptable appropriateness
Patient-defined qualitative appropriateness (Secondary Implementation) | Within 1 year of completing study procedures
  Themes from semi-structured interviews with patients related to intervention appropriateness will be identified
Provider-defined qualitative acceptability (Secondary Implementation) | Within 1 year of completing study procedures
  Themes from semi-structured interviews with providers related to intervention acceptability will be identified

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Corwin, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zemek R, Barrowman N, Freedman SB, Gravel J, Gagnon I, McGahern C, Aglipay M, Sangha G, Boutis K, Beer D, Craig W, Burns E, Farion KJ, Mikrogianakis A, Barlow K, Dubrovsky AS, Meeuwisse W, Gioia G, Meehan WP 3rd, Beauchamp MH, Kamil Y, Grool AM, Hoshizaki B, Anderson P, Brooks BL, Yeates KO, Vassilyadi M, Klassen T, Keightley M, Richer L, DeMatteo C, Osmond MH; Pediatric Emergency Research Canada (PERC) Concussion Team. Clinical Risk Score for Persistent Postconcussion Symptoms Among Children With Acute Concussion in the ED. JAMA. 2016 Mar 8;315(10):1014-25. doi: 10.1001/jama.2016.1203. PMID 26954410
- [Background] Corwin DJ, Arbogast KB, Haber RA, Pettijohn KW, Zonfrillo MR, Grady MF, Master CL. Characteristics and Outcomes for Delayed Diagnosis of Concussion in Pediatric Patients Presenting to the Emergency Department. J Emerg Med. 2020 Dec;59(6):795-804. doi: 10.1016/j.jemermed.2020.09.017. Epub 2020 Oct 7. PMID 33036827
- [Background] Master CL, Master SR, Wiebe DJ, Storey EP, Lockyer JE, Podolak OE, Grady MF. Vision and Vestibular System Dysfunction Predicts Prolonged Concussion Recovery in Children. Clin J Sport Med. 2018 Mar;28(2):139-145. doi: 10.1097/JSM.0000000000000507. PMID 29064869
- [Background] Desai N, Wiebe DJ, Corwin DJ, Lockyer JE, Grady MF, Master CL. Factors Affecting Recovery Trajectories in Pediatric Female Concussion. Clin J Sport Med. 2019 Sep;29(5):361-367. doi: 10.1097/JSM.0000000000000646. PMID 31460948
- [Background] Wiebe DJ, Nance ML, Houseknecht E, Grady MF, Otto N, Sandsmark DK, Master CL. Ecologic Momentary Assessment to Accomplish Real-Time Capture of Symptom Progression and the Physical and Cognitive Activities of Patients Daily Following Concussion. JAMA Pediatr. 2016 Nov 1;170(11):1108-1110. doi: 10.1001/jamapediatrics.2016.1979. No abstract available. PMID 27617669
- [Background] Corwin DJ, Orchinik J, D'Alonzo B, Agarwal AK, Pettijohn KW, Master CL, Wiebe DJ. A Randomized Trial of Incentivization to Maximize Retention for Real-Time Symptom and Activity Monitoring Using Ecological Momentary Assessment in Pediatric Concussion. Pediatr Emerg Care. 2023 Jul 1;39(7):488-494. doi: 10.1097/PEC.0000000000002870. Epub 2022 Nov 3. PMID 36730797
- [Derived] Corwin DJ, Godfrey M, Arbogast KB, Zorc JJ, Wiebe DJ, Michel JJ, Barnett I, Stenger KM, Calandra LM, Cobb J, Winston FK, Master CL. Using mobile health to expedite access to specialty care for youth presenting to the emergency department with concussion at highest risk of developing persisting symptoms: a protocol paper for a non-randomised hybrid implementation-effectiveness trial. BMJ Open. 2024 Jun 19;14(6):e082644. doi: 10.1136/bmjopen-2023-082644. PMID 38904136